CLINICAL TRIAL: NCT00789607
Title: Fiducial Localization and Individualized Radiotherapy in Prostate Cancer (FLIP)
Brief Title: Fiducial Localization and Individualized Radiotherapy -Prostate Cancer
Acronym: FLIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 08-0271-C
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; individualized radiotherapy; fiducial markers; MRI; ultrasound; High-Risk Localized Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MRI-guided FM (Active Comparator)
  Interventions: Device: Transrectal APT Device or Transperineal Device will be used
- TRUS-guided FM (Active Comparator)
  Interventions: Device: TRUS probe

INTERVENTIONS:
Device: Transrectal APT Device or Transperineal Device will be used — Both are imaging probe devices that is inserted under local anesthetic, in the rectum using lubricant, positioning against the prostate gland, and attached to the table. This is done at baseline (Day 0) under local anesthetic with the patient in partial dorsal lithotomy position
  Arms: MRI-guided FM
Device: TRUS probe — Patient is given local anesthetic transrectally to the prostate base and the probe is inserted with patient in the lateral decubitus position.
  Arms: TRUS-guided FM

SUMMARY:
This purpose of this study is designed to compare two types of images; magnetic resonance imaging (MRI) and Trans-Rectal Ultrasound (TRUS) to see which one performs more accurately for the image-guided insertion of Fiducial Markers(FMs) within the tumour. Though effective for guiding FM placement at the poles of the prostate gland due to excellent visualization of the prostatic boundaries, TRUS may not be ideally suited for marking the GTV. Conventional TRUS is neither sufficiently sensitive nor specific for accurate visualization of intra-prostatic tumor. A new interventional MRI technique enables needle guidance to the gross tumour Volume (GTV) for FM placement. It is of particular importance that both techniques be evaluated to enable which one is more effective so that it can be implemented in the designs of future trials involving dose-escalation to prostate.

DETAILED DESCRIPTION:
The success of dose escalation strategies in prostate cancer over the last decade has relied on high accuracy in target delineation, localization and radiation delivery. Improved biochemical control with acceptable levels of toxicity (specifically rectal) has been achieved by stringently monitoring the location of the prostate during the course of radiation treatment. Studies in the early 1990's demonstrated that daily bony alignment was a poor surrogate for prostate gland location. Since then, various strategies have been devised to localize the prostate precisely during treatment. Of these, Transrectal Ultrasound (TRUS)-guided gold fiducial marker (FM) insertion and x-ray imaging of markers has been a broadly successful approach. TRUS guidance has been used for fiducial marker insertion within the prostate since 1985 in various centers throughout the world and has also been a standard practice in PMH since 1997 in men undergoing radical external beam radiotherapy. A retrospective comparative study of 106 patients evaluating the relative accuracy of endorectal MRI and TRUS in detecting the location of tumor reported an improved performance of endorectal MRI especially in the base and midgland regions. Over the last few years, mounting experience in the interpretation of prostate MRI, and addition of physiologic imaging sequences has further improved the performance of MRI in detecting and localizing the GTV.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old
2. ECOG status ≤ 1
3. High risk localized cancer planned for RT under FM guidance
4. Gleason > 7, PSA > 20, Clinical stage ≥ T3
5. patients(pts) must give written informed consent

Exclusion Criteria:

1. pts > 136 kg or > 60 cm in girth
2. Pts with pacemakers, cerebral aneurysm clips, shrapnel injury or devices not compatible with MRI.
3. pts with severe claustrophobia
4. pts with bleeding diathesis and anticoagulative therapy that cannot be ceased prior to needle procedures.
5. Contraindications to endorectal probe, surgically absent rectum, severe hemorrhoids or previous colorectal surgery.
6. Latex Allergy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-06; Primary Completion 2017-06 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
To compare the performance of MRI and TRUS images in guiding the insertion of a fiducial marker within the Gross Target Volume (GTV) | 5 years

SECONDARY OUTCOMES:
To measure the needle targeting accuracy of the MRI-guided technique. | 5 years
To validate the accuracy of identifying the GTV on MRI. | 5 years
To evaluate MRI methods for the characterization of tissue oxygenation. | 5 years
To evaluate the effect of neoadjuvant hormone therapy on tissue oxygenation. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Chung, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada